CLINICAL TRIAL: NCT01934608
Title: A Randomized Controlled Trial to Test a Synchronized Prescription Refill Program to Improve Medication Adherence
Brief Title: The Effect of Synching Prescription Refills on Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM-001
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension; Hypercholesterolemia; Diabetes; Medication Adherence
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Refill synch (Experimental): Participants in this group will have their medication refill schedule synchronized.
  Interventions: Behavioral: Refill synch
- Control (No Intervention): Participants in this arm will receive usual care

INTERVENTIONS:
Behavioral: Refill synch
  Arms: Refill synch

SUMMARY:
To determine the effect of synchronizing a patient's prescription refill schedule on medication adherence. The targeted population is Humana members who are currently taking 2 or more Stars medications (hypertension, hypercholesterolemia, diabetes) and are current customers of RightSource. Participants will be randomized to one of two groups. Group one will be usual care and group two will be the Rx synchronization group.

ELIGIBILITY:
Inclusion Criteria:

* Humana members who are currently taking 2 or more Stars medications (hypertension, hypercholesterolemia, diabetes) and are current customers of RightSource.

Exclusion Criteria:

* under 18 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Medication adherence to each of the chronic medications as measured by the proportion of days covered (PDC) measure | 6 months and 12 months

SECONDARY OUTCOMES:
Secondary outcomes will be continuous gaps (e.g. 15, 30, or 60 days) in medication use. | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jalpa Doshi, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Humana, Inc, Louisville, Kentucky, United States